CLINICAL TRIAL: NCT04286438
Title: A Phase 3, Multicenter, Open-Label, Single-Arm Study of Bentracimab (PB2452) in Ticagrelor-Treated Patients With Uncontrolled Major or Life-Threatening Bleeding or Requiring Urgent Surgery or Invasive Procedure (REVERSE-IT Trial)
Brief Title: Bentracimab in Ticagrelor-treated Patients With Uncontrolled Bleeding or Requiring Urgent Surgery or Invasive Procedure
Acronym: REVERSE-IT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SFJ Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB2452-PT-CL-0004; 2019-004457-92 (EudraCT Number)
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Hemorrhage; Urgent Surgery; Invasive Procedure
Keywords: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — PB-2452

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bentracimab (PB2452) Infusion - Open Label Active Drug (Experimental): Bentracimab (PB2452) 18 g Intravenous Infusion over a 16 hour duration. For patients with uncontrolled major or life-threatening bleeding or in need of urgent surgery or invasive procedure.
  Interventions: Drug: Bentracimab (PB2452) Infusion

INTERVENTIONS:
Drug: Bentracimab (PB2452) Infusion — Bentracimab (PB2452) 18 g Intravenous Infusion over a 16 hour duration.
  In subjects with potential drug interaction from recent concomitant use of moderate or strong CYP3A inhibitors with ticagrelor, the active treatment period may be 24 hours and 10 min if receiving the 36g infusion.
  In patients presenting with intracranial hemorrhage (ICH), brain imaging within 2 hours of initiation of study drug and at least one follow-up brain imaging performed 12-24 hours post completion of PB2452.

SUMMARY:
This is a multi-center, open-label, prospective single-arm study of reversal of the antiplatelet effects of ticagrelor with bentracimab (PB2452) in patients who present with uncontrolled major or life-threatening bleeding or who require urgent surgery or invasive procedure.

At least 200 patients will be enrolled from approximately 200 centers in North America, Europe, and Asia-Pacific regions, including mainland China. Patients with reported use of ticagrelor within the prior 3 days who require urgent ticagrelor reversal will be eligible for enrollment. These populations will be enrolled based on separate inclusion criteria.

DETAILED DESCRIPTION:
The study will consist of a Screening/Pre-treatment period, an on-site assignment to study treatment and administration, a Follow-up visit on (Day 3+1 and Day 7±1), a Final Follow-up visit (Day 35±3) and a Follow-up visit for intracranial hemorrhage (ICH) only patients (Day 90±10). Infusion of PB2452 will be initiated on Day 1 and will continue for approximately 16 hours for a total of 18 g.

On Day 1, subjects who meet all the inclusion criteria and none of the exclusion criteria will receive an intravenous (IV) infusion comprised of an initial IV bolus of 6 grams (g) infused over 10 minutes for rapid reversal, followed immediately by a 6g IV loading infusion over 4 hours and then a 6 g IV maintenance infusion over 12 hours. This bentracimab (PB2452) regimen is expected to provide immediate reversal of the antiplatelet effects of ticagrelor within 5 minutes of the initiation of infusion that is sustained for 20-24 hours.

In subjects with potential drug interaction from recent concomitant use of moderate or strong CYP3A inhibitors with ticagrelor, an alternative regimen may be used comprising administration of 36 g over an active treatment period of 24 hours and 10 min. (This alternative regimen will be an initial 12 g bolus infusion over 10 minutes, followed immediately by a loading infusion of 12 g over 6 hours which will then be followed by a maintenance regimen of 12 g infused over 18 hours for a total infusion of 36 grams over 24 hours and 10 minutes).

In patients presenting with intracranial hemorrhage (ICH), brain imaging within 2 hours of initiation of study drug and at least one follow-up brain imaging performed 12-24 hours post completion of PB2452 will be required to support adjudication of hemostasis.

All subjects may be discharged from the clinical site between Days 3 and 7 inclusive and will return for a Follow-up visit on Day 7, if already discharged, and on Day 35 (± 3 days). All ICH patients must complete End of Study (EOS) Day 35±3 (Visit 5). ICH patients that agree to participate in the ICH-only-90-day-follow-up visit will have an additional visit on Day 90±10 (Visit 6).

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion into the study if they meet all of the following criteria:

1. Male or female >18 years of age with documented or verbal informed consent. Emergency consent may be obtained where permitted by local regulations and institutional approval.
2. History or documentation of ticagrelor intake within the prior 3 days
3. Patients described below who require urgent reversal of the antiplatelet effects of ticagrelor:

Patients with uncontrolled major or life-threatening bleeding, requiring urgent reversal of the antiplatelet effects of ticagrelor. It is expected that enrolled patients would have characteristics similar to those described below:

* Potentially life-threatening bleeding with signs or symptoms of hemodynamic compromise, e.g., systolic blood pressure < 90 mm Hg and signs or symptoms of low cardiac output not otherwise explained
* Bleeding in a critical organ or closed space, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular, pericardial, or intramuscular bleed with compartment syndrome
* Visible, uncontrolled bleeding associated with a corrected hemoglobin level < 8.0 g/dL, a fall in hemoglobin level of ≥ 2.0 g/dL (1.24 mmol/L) from a known baseline, or requirement for transfusion of 2 or more units of packed red blood cells (PRBC)

Patients requiring urgent surgery or invasive procedure when it is not medically advisable either to proceed urgently with impaired hemostasis or to delay the urgent procedure for 3 or more days due to the high risk of bleeding. These patients may typically be in any of the following clinical situations:

* Requires urgent surgery or invasive procedure known to be associated with a risk of significant bleeding (such as cardiac surgery, neurosurgery, or major orthopedic surgery)
* Requires urgent surgery or invasive procedure that may have an adverse procedural outcome if hemostasis is impaired (such as neurological, spinal, ophthalmological, urological, or orthopedic surgery)
* At risk of experiencing life-threatening events, such as, shock, myocardial infarction, or stroke, if significant intraoperative or postoperative bleeding occurs (such as in elderly patients or patients with underlying cardiac or pulmonary disease who have limited cardiopulmonary reserve)

Exclusion Criteria:

1. Known sensitivity or contraindication to PB2452 or any of its excipients
2. Patients in whom ticagrelor reversal is not considered urgent, e.g., patients with stable or non-acute conditions who have low hemoglobin due to chronic, low-grade gastrointestinal bleeding or who have stable, remote, or asymptomatic intracranial hemorrhage
3. Patients expected to be clinically unsalvageable, such as, patients with end-stage cancer or patients with overwhelming sepsis
4. Any condition which, in the opinion of the investigator, would make it unsafe or unsuitable for the patients to participate in this study. This includes assessment of likelihood to cooperate with study follow-up visits and procedures. Known pregnancy may be exclusionary in some regions or countries as directed by national health authorities and/or local Institutional Review Boards/Ethics Committees
5. Known use of clopidogrel, prasugrel or ticlopidine within 5 days of study drug administration; known use of antiplatelet GPIIb/IIIa inhibitors, or cangrelor within 5 half-lives of expected study drug administration; or known use of warfarin, dabigatran, rivaroxaban, apixaban, or edoxaban within 5 half-lives of expected study drug administration
6. Known recent use (< 5 day) of vitamin K, prothrombin complex concentrate, recombinant factor VIIa, idarucizumab, or andexanet-alfa (coagulation factor Xa (recombinant), inactivated-zhzo)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Reversal - Platelet Reactivity Units (PRU) | 4 hours post-initiation of infusion
  Minimum % inhibition of PRU within 4 hours of the initiation of study drug as assessed by VerifyNow™ PRUTest™ platelet function assay
Hemostasis - Uncontrolled major of life-threatening bleeding - Achievement | 4 hours post-initiation of infusion
  Achievement of effective (graded as good or excellent) hemostasis after initiation of PB2452 infusion will be assessed using prespecified criteria for effective hemostasis for visible and non-visible major bleeding [Scale (from best to worst) measured as: Excellent, Good, Poor/None]
Hemostasis - Urgent surgery or invasive procedure - Achievement | 4 hours post-initiation of infusion
  Achievement of effective hemostasis following initiation of PB2452 infusion will be centrally adjudicated using prespecified criteria for effective hemostasis derived from the Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) clinical bleeding scale [GUSTO scale (from best to worst): Effective (no bleeding, mild bleeding or moderate bleeding) or Not effective (severe bleeding)]

SECONDARY OUTCOMES:
Minimum % inhibition of Platelet Reactivity Index (PRI) (VASP) | 4 hours post-initiation of infusion
  Minimum % inhibition of PRI assessed by VASP within 4 hours after the initiation of study drug
Maximum reversal of PRU assessed by VerifyNow™ PRUTest™ | 4 hours post-initiation of infusion
  Maximum reversal of PRU assessed by VerifyNow™ PRUTest™ within 4 hours after the initiation of study drug.
Maximum reversal of PRI assessed by VASP | 4 hours post-initiation of infusion
  Maximum reversal of PRI assessed by VASP within 4 hours after the initiation of study drug.
Proportion of subjects achieving reversal of platelet inhibition of ticagrelor using PRU and PRI - 60% | Any time point between infusion initiation and Day 3 (Pre-dose, 5-10 minutes, 30+5 minutes, 1+0.25 hours, 4+0.25 hours, 12+0.5 hours, 24+1 hours, and Day 3)
  Proportion of subjects achieving 60% reversal of platelet inhibition by ticagrelor using PRU and PRI at any time point during the treatment period
Proportion of subjects achieving reversal of platelet inhibition of ticagrelor using PRU and PRI - 80% | Any time point between infusion initiation and Day 3 (Pre-dose, 5-10 minutes, 30+5 minutes, 1+0.25 hours, 4+0.25 hours, 12+0.5 hours, 24+1 hours, and Day 3)
  Proportion of subjects achieving 80% reversal of platelet inhibition by ticagrelor using PRU and PRI at any time point during the treatment period
Proportion of subjects achieving reversal of platelet inhibition of ticagrelor using PRU and PRI - 100% | Any time point between infusion initiation and Day 3 (Pre-dose, 5-10 minutes, 30+5 minutes, 1+0.25 hours, 4+0.25 hours, 12+0.5 hours, 24+1 hours, and Day 3)
  Proportion of subjects achieving 100% reversal of platelet inhibition by ticagrelor using PRU and PRI at any time point during the treatment period
Duration of at least 60% reversal by PRU and PRI | Any time point between infusion initiation and Day 3 (Pre-dose, 5-10 minutes, 30+5 minutes, 1+0.25 hours, 4+0.25 hours, 12+0.5 hours, 24+1 hours, and Day 3)
Duration of at least 80% reversal by PRU and PRI | Any time point between infusion initiation and Day 3 (Pre-dose, 5-10 minutes, 30+5 minutes, 1+0.25 hours, 4+0.25 hours, 12+0.5 hours, 24+1 hours, and Day 3)
Duration of at least 100% reversal by PRU and PRI | Any time point between infusion initiation and Day 3 (Pre-dose, 5-10 minutes, 30+5 minutes, 1+0.25 hours, 4+0.25 hours, 12+0.5 hours, 24+1 hours, and Day 3)
Intracranial hemorrhage (ICH) Patients Only: Proportion of ICH patients with modified Rankin Scale (mRS) score of 0-3 versus 4-6 at 90 days on a scale of 0-6 (better to worse) | [Time Frame: Pre-dose, Day 35 and Day 90]
ICH Patients Only: Absolute and percent change form baseline in modified Rankin Scale (mRS) score at 90 days in ICH patients on a scale of 0-6 (better to worse) | [Time Frame: Pre-dose, Day 35 and Day 90]
ICH Patients Only: EQ-5D 5L Quality of Life Questionnaire index at 90 days and change from baseline in ICH patients on a scale of 0-100 (best to worst) | [Time Frame: Pre-dose, Day 35 and Day 90]

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Bhatt, MD, MPH, Study Chair — Brigham and Women's Hospital, Division of Cardiovascular Medicine
Locations (68):
- United States (9):
  - University of Florida Health, Jacksonville, Jacksonville, Florida
  - University of Kentucky, Lexington, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - North Kansas City Hospital, North Kansas City, Missouri
  - Cox Medical Centers, Springfield, Missouri
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Ascension St. John Clinical Research Institute, Tulsa, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
- Austria (3):
  - Medical University Of Graz, Graz, STY
  - Klinische Abteilung für Innere Medizin 3 Universitätsklinikum St. Pölten, Sankt Pölten
  - Klinik Ottakring 3rd Med Dept, Cardiology and Intensive Care Medicine, Vienna
- Belgium (5):
  - Algemeen Stedelijk Ziekenhuis (ASZ) Study Center Cardiology, Aalst, East Flanders
  - Ziekenhuis Oost-Limburg Study Center Intensive Care, Genk, Limburg
  - AZ Sint-Jan Brugge-Oostende AV Poli Cardiologie, Bruges
  - University Hospital Antwerp Cardiology Department - Clinical Trials, Edegem
  - Jessa Hospital Hartcentrum Hasselt Research Center, Hasselt
- Canada (9):
  - Foothills Medical Centre, Calgary, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - William Osler Health System, Etobicoke, Ontario
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston Health Science Centre, Kingston, Ontario
  - York PCI Group, Inc., Newmarket, Ontario
  - St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
- China (21):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Medidata, Hangzhou, Zhejiang
  - Shanghai General Hospital, Shanghai
- France (4):
  - CHU de Lille Service USIC, Institut Coeur Poumon, Lille
  - Assistance Publique-Hopitaux de Paris (AP-HP) Pitie-Salpetriere Hospital, Paris
  - Bichat Hospital, Service de Cardiologie, Paris
  - CHRU de Tours - Hopital Trousseau Service de Cardiologie-USCI 2 eme etage, Tours
- Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen, Germany
- Italy (3):
  - ASST Monza - Ospedale San Gerardo, Monza
  - Azienda Ospedaliero-Universitaria di Parma Cardiologia, Parma
  - Istituto Clinico Humanitas UO Cardiologia Clinica e Interventistica, Rozzano
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede, Overijssel
  - St Antonius Hospital, Nieuwegein
- Spain (5):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Residencia general, Madrid
  - Hospital Universitario Vírgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Department of Cardiology, Lund
- Switzerland (2):
  - Universitatsspital Basel Department of Cardiology, Basel
  - Cardiocentro Ticino, Lugano
- United Kingdom (2):
  - East and North Hertfordshire, NHS Trust, Lister Cardiac Research Office, Cardiology Green Zone, Lister Hospital, Stevenage, Hertfordshire
  - Sheffield Teaching Hospitals, NHS Foundation Trust, Northern General Hospital, Sheffield

REFERENCES:
- [Derived] Bhatt DL, Pollack CV, Mazer CD, Angiolillo DJ, Steg PG, James SK, Weitz JI, Ramnath R, Arnold SE, Mays MC, Umstead BR, White B, Hickey LL, Jennings LK, Curry BJ, Lee JS, Verma S. Bentracimab for Ticagrelor Reversal in Patients Undergoing Urgent Surgery. NEJM Evid. 2022 Mar;1(3):EVIDoa2100047. doi: 10.1056/EVIDoa2100047. Epub 2021 Dec 1. PMID 38319214